CLINICAL TRIAL: NCT02100839
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of AEM-28 in Healthy Subjects and Patients With Refractory Hypercholesterolemia
Brief Title: Safety Study of AEM-28 to Treat Refractory Hypercholesterolemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LipimetiX Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPMX-112
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-03

CONDITIONS: Hypercholesterolemia; Hyperlipoproteinemia Type II
Keywords: hypercholesterolemia; apolipoprotein E; First in Human; Apolipoprotein E (ApoE); Apolipoprotein E Mimetic (AEM)
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — apolipoprotein E mimetic peptide CN-105; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AEM-28 (Experimental): Single Ascending Dose: Single IV dose for each cohort; dose range 0.032 mg/mL to 3.54 mg/mL
  Multiple Ascending Dose: Three (3) IV doses for each cohort, one (1) dose every two (2) weeks; dose range 1 mg/kg to 3.54 mg/kg.
  Interventions: Drug: AEM-28
- Normal Saline (Placebo Comparator): Single Ascending Dose: Single IV dose for each cohort.
  Multiple Ascending Dose: Three (3) IV doses for each cohort, one (1) dose every two (2) weeks.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: AEM-28 — Solution for injection
  Other Names: apolipoprotein E mimetic
  Arms: AEM-28
Drug: Normal Saline — 0.9% saline for injection
  Other Names: 0.9% NaCl; Sterile Normal Saline
  Arms: Normal Saline

SUMMARY:
The purpose of the first part of this study is to determine the safety and tolerability of a single dose of AEM-28, an apolipoprotein E mimetic, in subjects with high total cholesterol who are otherwise healthy subjects. The pharmacokinetics and pharmacodynamics of AEM-28 will also be evaluated.

The second part of this study will be a multiple ascending dose evaluation of AEM-28 in patients with refractory hypercholesterolemia.

AEM-28 has demonstrated significant lipid lowering activity and positive effects on the artery wall. AEM-28 is being developed for the treatment of homozygous familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

Single Ascending Dose (SAD) Study:

* Male or female non-smoker, ≥18 and ≤55 years of age, with BMI >18.5 and < 32.0 kg/m²
* Total cholesterol greater or equal to 5.0 mmol/L (≥194 mg/dL) at screening

Multiple Ascending Dose (MAD) Study:

* Male or female non-smoker, ≥18 and ≤75 years of age, with BMI >18.5 and < 35.0 kg/m²
* Diagnosis of refractory hypercholesterolemia with LDL cholesterol levels > 2.5 mmol/L (97 mg/mL) at screening.
* On stable lipid lowering therapy for ≥ 8 weeks
* On stable diet for ≥ 12 weeks.

Exclusion Criteria:

SAD Study:

* Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
* History of allergic reactions to diphenhydramine, ranitidine, methylprednisone or other related drugs, or history of significant allergic or hypersensitivity reaction (e.g. angioedema) to any substance.

MAD Study:

* Significant health problems within 6 months prior to screening, which in the opinion of the Medical Sub-Investigator would prevent the subject from participating in the study, including but not limited to: unstable coronary heart disease; transient ischemic attack; stroke; revascularization procedure; uncontrolled hyperthyroidism; coagulation disorder; peptic ulcers or GI bleeding; significant disease of the central nervous system; liver or renal disease.
* History of allergic reactions to diphenhydramine, ranitidine, methylprednisone or other related drugs, or history of significant allergic or hypersensitivity reaction (e.g. angioedema) to any substance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janakan Krishnarajah, MBBS, FRACP, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research Ltd., Nedlands, Western Australia, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted at Linear Clinical Research Ltd, a medical clinic in Nedlands WA Australia.
Groups:
- Apolipoprotein E Mimetic (AEM)-28: Single Ascending Dose (SAD): Single IV dose for each cohort; dose range 0.032 mg/mL to 3.54 mg/mL
  Multiple Ascending Dose (MAD): Three (3) IV doses for each cohort, one (1) dose every two (2) weeks; dose range 1 mg/kg to 3.54 mg/kg.
  AEM-28: Solution for injection
- Normal Saline: Single Ascending Dose: Single IV dose for each cohort.
  Multiple Ascending Dose: Three (3) IV doses for each cohort, one (1) dose every two (2) weeks.
  Normal Saline: 0.9% saline for injection
Period: Single Ascending Dose
Arm/Group | Apolipoprotein E Mimetic (AEM)-28 | Normal Saline
Started | 24 | 12
Completed | 24 | 12
Not Completed | 0 | 0
Period: Multiple Ascending Dose
Arm/Group | Apolipoprotein E Mimetic (AEM)-28 | Normal Saline
Started | 13 | 3
Completed | 9 | 3
Not Completed | 4 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- AEM-28: Single Ascending Dose: Single IV dose for each cohort; dose range 0.032 mg/mL to 3.54 mg/mL
  Multiple Ascending Dose: Three (3) IV doses for each cohort, one (1) dose every two (2) weeks; dose range 1 mg/kg to 3.54 mg/kg.
  AEM-28: Solution for injection
- Total: Total of all reporting groups
Arm/Group | AEM-28 | Normal Saline | Total
Number analyzed (Participants) | 37 | 15 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 15 | 50
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 35.7 [18 to 67] | 32 [18 to 48] | 34.6 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 30 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 33 | 15 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 31 | 11 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Australia | 37 | 15 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Incurred at Least One Treatment Emergent Event
Description: Safety and tolerability to AEM-28 were evaluated through the assessment of adverse events (i.e., seriousness, severity, relationship to the study medication, outcome, duration, and management), vital signs, 12-lead ECG, telemetry, clinical laboratory parameters, physical examination, and local response to each injection, and body weight (Part B only). Treatment-emergent adverse events were tabulated by treatment. Changes from baseline values in vital signs, ECG, clinical laboratory parameters, physical examination, and body weight (Part B only) were evaluated.
  Safety and tolerability data were reported using descriptive statistics.
Time Frame: Part A (SAD): Day -1 to Day 15; Part B (MAD): Day 1 to Day 57
Measure: Number; unit: participants
Arm/Group | AEM-28 | Normal Saline
Number analyzed (Participants) | 37 | 15
participants | 33 | 10

2. Primary Outcome: Number of Participants Who Incurred Mild Treatment Emergent Adverse Events
Description: as for outcome 1
Time Frame: Part A (SAD): Day -1 to Day 15; Part B (MAD): Day 1 to Day 57
Measure: Number; unit: Number of Participants
Arm/Group | AEM-28 | Normal Saline
Number analyzed (Participants) | 37 | 15
Number of Participants | 33 | 10

3. Primary Outcome: Number of Participants Who Incurred Moderate Treatment Emergent Events
Description: as for outcome 1
Time Frame: Part A (SAD): Day -1 to Day 15; Part B (MAD): Day 1 to Day 57
Measure: Number; unit: Number of Participants
Arm/Group | AEM-28 | Normal Saline
Number analyzed (Participants) | 37 | 15
Number of Participants | 7 | 0

4. Secondary Outcome: Very Low Density Lipoprotein Cholesterol (VLDL-C) Percent Change
Description: Maximum observed percentage change in VLDL-C level relative to baseline for all time points measured in Parts A or Part B with highest dose, i.e. 3.54 mg/kg.
Time Frame: Part A (SAD): Day 1 to Day 15; Part B (MAD): Day 1 to Day 57
Measure: Mean (Standard Deviation); unit: Max % Change Versus Baseline
Arm/Group | AEM-28 | Normal Saline
Number analyzed (Participants) | 37 | 15
Max % Change Versus Baseline
  Part A: 3.54 mg/kg | -72.1 (15.1) | -0.33 (0.17)
  Part B: 3.54 mg/kg | -79.2 (13.5) | -0.58 (0.31)
  Part A: 2.0 mg/kg | -76.3 (7.25) | -0.35 (0.13)
  Part B: 2.0 mg/kg | -73.3 (6.36) | -0.52 (0.15)
  Part A: 1.0 mg/kg | -47.9 (19.7) | -0.23 (0.15)
  Part B: 1.0 mg/kg | -51.8 (24.7) | -0.38 (0.19)

ADVERSE EVENTS:
Time Frame: Over 8 day study period for SAD study, and over 57 day study period for MAD study
Arm/Group | AEM-28 | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/15
Other Adverse Events (participants affected / at risk) | 33/37 | 10/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEM-28 (N=37) | Normal Saline (N=15)
Administration Site Reaction (General disorders) | 29 (46) | 6 (7) — Infusion site bruising, erythema, pain, phlebitis, swelling
Headache (Nervous system disorders) | 9 (12) | 0 (0)
Confusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 6 (13) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No